CLINICAL TRIAL: NCT04995159
Title: Evaluate the Safety and Efficacy of Optimized Antiplatelet Therapy in Patients With Coronary Heart Disease After Implantation of NeoVas™ Bioabsorbable Coronary Artery Rapamycin-eluting Stent System.
Brief Title: Optimized Antiplatelet Therapy in Patients With CHD After Implantation of NeoVas™ BRS System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPT-BRS
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Coronary Heart Disease
Keywords: Bioabsorbable Coronary Artery Rapamycin-eluting Stent System; Optimized Antiplatelet Therapy; Coronary Heart Disease; Randomized Controlled Trial
MeSH Terms: conditions — Coronary Disease | interventions — Dual Anti-Platelet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Poststent SAPT treatment cohort (Experimental): receiving the treatment with NeoVas™ Bioabsorbable Coronary Artery Rapamycin-eluting Stent System of Lepu Medical combined with SAPT strategy
  Interventions: Drug: Single anti-platelet therapy
- Poststent DAPT treatment cohort (Active Comparator): receiving the treatment with NeoVas™ Bioabsorbable Coronary Artery Rapamycin-eluting Stent System of Lepu Medical combined with DAPT strategy
  Interventions: Drug: Dual anti-platelet therapy

INTERVENTIONS:
Drug: Single anti-platelet therapy — Aspirin in combination with a P2Y12 receptor antagonist (either clopidogrel or ticagrelor will be selected by investigators according to the degree of ischemia) in the first year after PCI. Aspirin will be discontinued one year after surgery and clopidogrel will be continued until 5 years after surgery.
  Other Names: SAPT strategy
  Arms: Poststent SAPT treatment cohort
Drug: Dual anti-platelet therapy — Aspirin in combination with a P2Y12 receptor antagonist (either clopidogrel or ticagrelor will be selected by investigators according to the degree of ischemia) in the first year after PCI. Patients continue to take dual antiplatelet (DAPT) drugs, including aspirin and clopidogrel, for 2 more years; then aspirin will be used alone from the 4th year to the 5th year.
  Other Names: DAPT strategy
  Arms: Poststent DAPT treatment cohort

SUMMARY:
This study is designed to verify the safety and efficacy of Lepu® NeoVas™ Bioabsorbable Coronary Artery Rapamycin-eluting Stent System combined with different antiplatelet therapies in the treatment of coronary heart disease.

DETAILED DESCRIPTION:
A total of 2150 subjects are planned to be enrolled in this trial. Subjects meeting the inclusion criteria and without exclusion criteria are implanted with NeoVas™ stents and randomly assigned to the experimental group and the control group in a 1:1 ratio. Patients in both groups will receive aspirin in combination with a P2Y12 receptor antagonist in the first year after PCI (either clopidogrel or ticagrelor will be selected by investigators according to the degree of ischemia). Aspirin will be discontinued one year after surgery and clopidogrel will be continued until 5 years after surgery in the experimental group. The control group will continue to take dual antiplatelet (DAPT) drugs, including aspirin and clopidogrel, for 2 more years; then aspirin will be used alone from the 4th year to the 5th year.

Subjects will be followed up at 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years after surgery to observe whether the net adverse clinical events (NACEs) and other end points occur or not.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above, male or non-pregnant female.
* Evidence of myocardial ischemia (e.g., stable angina, unstable angina, medium-low risk NSTEMI, STEMI with onset more than 1 week, old myocardial infarction or asymptomatic myocardial ischemia), and suitable for PCI surgery.
* The target lesion is in-situ coronary artery lesion, the total length of single lesion is no more than 40mm (the total length of stent is no more than 48mm), and the diameter of the target lesion is between 2.75mm and 3.75mm (visual measurement).
* The diameter stenosis of target lesion is ≥70% in visual (or ≥50% with clinical evidence of myocardial ischemia in that range), and the TIMI blood flow is greater than grade 1.
* The stent with diameter more than 3.0mm is allowed to overlap with another stent once, the overlapping methods could be edge to edge or at most 1mm overlap. The total number of stents per patient is no more than 4, with a maximum of 2 stents per vessel (the 2.75mm diameter stent is not allowed to overlap).
* Patient with indications for coronary artery bypass surgery.
* Aspirin and clopidogrel could be used continuously during the study.
* Patient who can understand the purpose of this trial, is willing to participate in the trial and to conduct clinical follow-up as required by the study protocol.

Exclusion Criteria:

* Acute ST-segment elevation myocardial infarction within 1 week.
* Left main coronary artery disease, branch vessel diameter≥2.0mm, three-vessel coronary artery disease and bridge vessel disease; visible thrombus in the target vessel.
* Severe distortion, severe calcification that cannot be successfully predilated, and other lesions that are not suitable for stent delivery and deployment.
* Intra-stent restenosis.
* Severe heart failure (NYHA≥III or left ventricular ejection fraction<35%).
* Severe renal insufficiency, eGFR<30ml/min/1.73m2 or serum creatinine>2.5mg/dL (221μmol/L).
* Patients with bleeding tendency, active gastrointestinal ulcer, history of cerebral hemorrhage or subarachnoid hemorrhage, history of stroke within half a year, fundus hemorrhage affecting vision, antiplatelet agents and anticoagulant treatment contraindications who cannot receive antithrombotic therapy.
* Patients requiring long-term oral anticoagulants during the study period.
* Patients who are pregnant, breastfeeding, or planning to become pregnant during the study period.
* Patients with malignancies, organ transplants, or drug addiction that can seriously affect study compliance.
* Patients with contraindications to aspirin, clopidogrel or ticagrelor.
* Known allergy to aspirin, clopidogrel, ticagrelor, heparin, contrast agent, polylactic acid polymer and rapamycin.
* Thrombosis occurred during previous clopidogrel treatment.
* Life expectancy is less than 36 months.
* Participated in clinical trials of other drugs or medical devices before enrollment and failed to meet the time limit of the primary end point.
* Patients who will have elective surgery within a year and need to discontinue aspirin, clopidogrel or ticagrelor.
* Subjects are deemed unsuitable for enrollment by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2150 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical event (NACE) | 3 years
  NACE includes POCE (including all-cause death, all non-fatal myocardial infarction (Universal Definition of Myocardial Infarction, 4th Edition), any revascularization, and stroke), and major bleeding events of grade 2, 3, and 5 as defined by BARC.

SECONDARY OUTCOMES:
Target lesion failure (TLF) | 3 years
  Target lesion failure (TLF) includes cardiac death, target vessel myocardial infarction (TV-MI) and ischemic-driven target lesion revascularization (ID-TLR).
Comparison of net adverse clinical events | 30 days, 6 months, 1 year, 2 years, 4 years, and 5 years
Bleeding events of grade 3 and 5 as defined by BARC | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
Bleeding events of grade 2, 3 and 5 as defined by BARC | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
Bleeding events of grade 1, 2, 3 and 5 as defined by BARC | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
Comparison of target lesion failures | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
Patient-oriented composite endpoint (PoCE) | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
  Patient-oriented composite endpoint (PoCE) includes all-cause death, all MI, any revascularization, and stroke.
Ischemic-driven target lesion revascularization (iTLR) | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
Ischemic-driven target vessel revascularization (iTVR) | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
All cardiac revascularization | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
  All cardiac revascularization includes PCI and CABG.
Two types of stent thrombosis events as defined by BRS_ARC2 | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Study Chair — The General Hospital of Northern Theater Command
Locations (114):
- China (114):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital with Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Capital Medical University-12 Ward, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Capital Medical University-28 Ward, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Capital Medical University-33 Ward, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuan Wu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Jingmei Group General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Foshan First People's Hospital, Foshan, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangdong Medical University, Guangzhou, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shenzhen University General Hospital, Shenzhen, Guangdong
  - Zhanjiang Central People's Hospital, Zhanjiang, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Guilin People's Hospital, Guilin, Guangxi
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First People's Hospital of Nanning, Nanning, Guangxi
  - Yulin First People's Hospital, Yulin, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Haikou People's Hospital, Haikou, Hainan
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Sanya Central Hospital (Hainan Third People's Hospital), Sanya, Hainan
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hengshui People's Hospital, Hengshui, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - the 980th Hospital of Chinese People's Liberation Army Joint Logistics Support Force, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Nanyang Central Hospital, Nanyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - The Second Affiliated Hospital, Zhengzhou University, Zhengzhou, Henan
  - The 7th People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Zhengzhou, Henan
  - The First Affiliated Hospital, Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Fifth Hospital in Wuhan, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science, Baotou, Inner Mongolia
  - Gynecology of Huai'an First People's Hospital, Nanjing Medical University, Huai'an, Jiangsu
  - Affiliated Lianyungang Hospital of Nanjing University of Chinese Medicine, Lianyungang, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Xuzhou Cancer Hospital, Xuzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Gannan Medical College, Ganzhou, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Yingtan People's Hospital, Yingtan, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Dalian Municipal Central Hospital Affiliated of Dalian Medical University, Dalian, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital Affiliated to School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality
  - Baoji Central Hospital, Baoji, Shanxi
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - First Affiliated Hospital of the Fourth Military Medical University, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Shanxi Provincial Hospital, Xi’an, Shanxi
  - Tangdu Hospital of the Fourth Military Medical University of the PLA, Yanan, Shanxi
  - Yan'an University Affiliated Hospital, Yanan, Shanxi
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Teda International Cardiovascular Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Fuwai Yunnan Cardiovascular Hospital, Kunming, Yunnan
  - The First People's Hospital of Yunnan, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang